CLINICAL TRIAL: NCT02493725
Title: A PROSPECTIVE, MULTI-CENTER, PHASE II STUDY TO EVALUATE THE SAFETY AND EFFICACY OF ECULIZUMAB IN SUBJECTS WITH GUILLAIN-BARRÉ SYNDROME
Brief Title: JET-GBS - Japanese Eculizumab Trial for GBS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chiba University (Other)
Collaborators: Japan Agency for Medical Research and Development (Other Government)
Responsible Party: Principal Investigator, Satoshi Kuwabara, Professor, Chiba University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 100069
Record Dates: First submitted 2015-07-07; First posted 2015-07-09 (Estimated); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: Gullain Barre Syndrome
MeSH Terms: interventions — eculizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Eculizumab (Active Comparator): Eculizumab, 900 mg intravenously once a week
  Interventions: Drug: Eculizumab
- Placebo (Placebo Comparator): Matched placebo, intravenously once a week
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eculizumab
  Arms: Eculizumab
Drug: Placebo
  Arms: Placebo

SUMMARY:
Guillain-Barré syndrome (GBS) is an immune-mediated polyneuropathy that usually follows an antecedent infection and causes acute neuromuscular paralysis. GBS is currently classified into the two major subtypes: a classical demyelinating type and axonal variant type. Whereas in Europe and North America demyelinating GBS is the major subtype, in East Asia and Central and South America, axonal GBS is found in 30~65% of patients. Although the pathophysiology of GBS has not been fully understood, major advances have been made in understanding the pathophysiology particularly for the axonal form of GBS. It is now established that axonal GBS is caused by molecular mimicry of human gangliosides by the Campylobacter jejuni lipo-oligosaccharides. Autoantibodies bind to GM1 or GD1a at the nodes of Ranvier, activate complements, and disrupt sodium channel clusters and axo-glial junctions, resulting in the nerve conduction failure and muscle weakness. C. jejuni infection induces production of antibodies, which cross-react with gangliosides on the human nerve axolemma, and activate the complements, resulting in formation of membrane attack complex (MAC). The pathology leads to axonal degeneration.

The standard treatments for GBS are plasma exchange and intravenous immunoglobulin and the disease progression reaches its nadir within 4 weeks. However, during the acute phase, 18-28 % of the patients require artificial ventilation and 4.1-6.3 % of the patients die of complications. Recovery takes several months or years, and 16.7-19.7 % of the patients still require aid to walk one year after onset. Because of such serious disability of GBS patients, an alternative novel therapy that can prevent death during acute phase or severe sequelae is needed.

Eculizumab is a humanized monoclonal antibody of murine anti-human C5 antibody and specifically binds to the final activation complement component C5 and inhibits MAC formation by suppressing the cleavage reaction of C5 into C5a and C5b. The efficacy of eculizumab against GBS has been shown in a model of axonal GBS. At present, there are no animal models of demyelinating GBS. However, autopsy studies have shown that C3d and C5b-9 (MAC) are deposited on the Schwan cells, and therefore eculizumab can be effective also for demyelinating GBS.

This clinical trial will be conducted to investigate the efficacy and safety of eculizumab for GBS to warrant future global clinical trials. Moreover, we also study the relationship between the efficacy and clinical subtypes of GBS, such as axonal or demyelinating form. Our trial will provide insights on whether the future global developmental plan should target the whole spectrum of GBS world-wide or focusing on Asia and South America.

ELIGIBILITY:
* Patients who have been diagnosed with GBS with reference to GBS NINDS(National Institute of Neurological Disorders and Stroke) diagnostic criteria and those who meet all the following inclusion criteria and do not fall under any of the exclusion criteria will be included in this trial.

Inclusion Criteria：

1. Subjects ≥ 18 years of age at the time of obtaining informed consent.
2. Patients with onset of muscular weakness due to GBS less than 2 weeks before the time of consent.
3. Patients unable to walk unaided for ≥5 meters (progressively deteriorating FG(Functional Grade)3 or FG 4-5).
4. Patients who are already on IVIg or deemed eligible for and who will start IVIg (Generally, administration of 400mg/kg over 5 days).
5. Patients who can start their first dose of eculizumab within 2 weeks from onset of weakness and before the end of the IVIg treatment period.
6. Female subjects of child bearing potential with a negative result in their pregnancy test. All subjects must be able to practice an effective, reliable, medically approved method of contraception during the IP(Intraperitoneal) administration period and up to 5 months after IP administration is ended.
7. Patients who can be hospitalized during IP administration period.
8. Patients who have signed the informed consent form.

Exclusion Criteria:

1. Patients who are being considered for or are already on plasmapheresis.
2. Patients who are pregnant or lactating.
3. Patients showing clear clinical evidence of peripheral polyneuropathy other than GBS, e.g. diabetic (except for mild sensory disturbance) or severe vitamin B1 deficiency related.
4. Patients who have received immunosuppressive treatment (e.g. azathioprine, cyclosporine, tacrolimus, or >20 mg prednisolone daily) during the 4 weeks prior to providing consent.
5. Patients who are known to have severe concurrent disease (such as malignancy with uncontrolled primary tumors or metastatic lesions, severe cardiovascular disease, severe COPD(chronic obstructive pulmonary disease ), or TB).
6. Patients who are unable to comply with study procedures and the treatment regimen.
7. Patients who have received rituximab within 24 weeks prior to providing consent.
8. Patients with a history of or unresolved Neisseria meningitides.
9. Patients with active infectious diseases determined to be clinically severe by the principal investigator or sub-investigator that are not being appropriately treated with antibiotics.
10. Patients who that cannot be treated with antibiotic prophylaxis due to allergies.
11. Patients who are allergic to eculizumab.
12. Patients who are known to have or are suspected of having hereditary complement deficiencies.
13. Patients who have been administered another investigational product within 12 weeks prior to providing consent or are currently participating in another trial.
14. Patients with any condition that, in the opinion of the principal investigator or sub-investigator, could increase the patient's risk by participating in the study or confound the outcome of the study.
15. Patients who have a history of Eculizumab treatment for GBS.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-07; Primary Completion 2016-05 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
[Safety] Expressed frequency and severity of incidence of AE/SAEs after treatment with investigational product. | 6 months
[Efficacy] Proportion of subjects who reach a score of FG2 or lower on the Hughes functional grading scale at week 4（Response Rate） | 4 weeks

SECONDARY OUTCOMES:
Proportion of subjects with improvement of one or more scores on the functional grading scale at each visit | 6 months
Proportion of subjects who are able to walk unaided (FG2 or lower) at each visit | 6 months
Duration required for improvement by at least one grade on the Hughes functional grading scale | 6 months
Proportion of subjects who reach FG1 or 0 at week 24 | 6 months
Change in the FG score between peak disability score and the scores at each visit | 6 months
Proportion of subjects with a clinically relevant improvement in the R-ODS score. An increase in the R-ODS score (0-48) converted to the centile metric score (0-100) by at least six points at each visit | 6 months
Proportion of subjects with a clinically relevant improvement in ONLS. (a decrease in the ONLS score from baseline by at least 1 point) at each visit | 6months
Proportion and frequency of subjects who require ventilatory support (F 5) | 4 weeks
Duration of ventilatory support | 8 weeks
Occurrence of relapse from the start of the IP(Investigational Product) administration period until the end of the post IP period | 2 years
Overall survival from the start of the IP administration period until the end of the post IP period (OS) | 6 months
Change in grip strength at each visit from baseline | 6 months
Change in results of the manual muscle test (MMT score) at each visit from baseline | 6 months
Change in the rate and results of below measures on the nerve conduction test parameter from baseline:Median and ulnar nerve 's CMAP amplitude, distal latency, F wave latency , SNAP amplitude, motor sensory nerve conduction velocity | 6 months
Change in vital capacity and % vital capacity at each visit from baseline | 6 months
Proportion of patients who undergo re-administration of IVIg | 6 months

OTHER OUTCOMES:
Antiganglioside antibodies (Antibodies to GM1・GD1a・GalNAc-GD1a・GQ1b, and their complexes) | 6 months
Concentration of eculizumab in serum | 6 months
Hemolytic complement activity in serum | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Satoshi Kuwabara, MD, Principal Investigator — Chiba University Graduate School of Medicine Department of neurology
Locations (13):
- Japan (13):
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - Kitasato University Hospital, Sagamihara, Kanagawa
  - Kindai University Hospital, Ōsaka-sayama, Osaka
  - National Defence Medical College Hospital, Tokorozawa, Saitama
  - Dokkyo Medical University Hospital, Mibu, Tochigi
  - Tokyo Medical and Dental University Hospital, Bunkyo-ku, Tokyo
  - Tokyo University Hospital, Bunkyo-ku, Tokyo
  - Keio University Hospital, Shinjuku-ku, Tokyo
  - Chiba University Hospital, Chiba
  - Kyushu University Hospital, Fukuoka
  - Tokushima University Hospital, Tokushima

REFERENCES:
- [Derived] Misawa S, Kuwabara S, Sato Y, Yamaguchi N, Nagashima K, Katayama K, Sekiguchi Y, Iwai Y, Amino H, Suichi T, Yokota T, Nishida Y, Kanouchi T, Kohara N, Kawamoto M, Ishii J, Kuwahara M, Suzuki H, Hirata K, Kokubun N, Masuda R, Kaneko J, Yabe I, Sasaki H, Kaida KI, Takazaki H, Suzuki N, Suzuki S, Nodera H, Matsui N, Tsuji S, Koike H, Yamasaki R, Kusunoki S; Japanese Eculizumab Trial for GBS (JET-GBS) Study Group. Safety and efficacy of eculizumab in Guillain-Barre syndrome: a multicentre, double-blind, randomised phase 2 trial. Lancet Neurol. 2018 Jun;17(6):519-529. doi: 10.1016/S1474-4422(18)30114-5. Epub 2018 Apr 21. PMID 29685815
- [Derived] Yamaguchi N, Misawa S, Sato Y, Nagashima K, Katayama K, Sekiguchi Y, Iwai Y, Amino H, Suichi T, Yokota T, Nishida Y, Kohara N, Hirata K, Nishiyama K, Yabe I, Kaida KI, Suzuki N, Nodera H, Tsuji S, Koike H, Kira JI, Hanaoka H, Kusunoki S, Kuwabara S; JET-GBS Group. A Prospective, Multicenter, Randomized Phase II Study to Evaluate the Efficacy and Safety of Eculizumab in Patients with Guillain-Barre Syndrome (GBS): Protocol of Japanese Eculizumab Trial for GBS (JET-GBS). JMIR Res Protoc. 2016 Nov 7;5(4):e210. doi: 10.2196/resprot.6610. PMID 27821382